CLINICAL TRIAL: NCT04255030
Title: An Adaptive Dyadic Self-directed Coping and Self-management Skills Training Intervention for Caregivers of Individuals With Cancer: A Pilot Sequential Multiple Assignment Randomized Trial (SMART) Design
Brief Title: An Adaptive Dyadic Self-directed Coping and Self-management Skills Training Intervention for Caregivers of Individuals With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Sylvie Lambert, Principal Scientist, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMHC 17 10
Record Dates: First submitted 2019-11-01; First posted 2020-02-05 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cancer; Anxiety
Keywords: Caregiver; Self-directed interventions; Coping; Self-management; Stepped care; Psychosocial oncology; Cancer; Sequential Multiple Assignment Randomized Trial (SMART)
MeSH Terms: conditions — Neoplasms; Anxiety Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First stage: Self-directed Coping Together (Experimental)
  Interventions: Behavioral: Coping Together Booklets and Workbook
- First stage: Minimally guided telephone support (lay coaching) (Experimental)
  Interventions: Behavioral: Coping Together Booklets and Workbook; Behavioral: Lay telephone coaching
- Second stage: High intensity Motivational Interviewing (MI) (Experimental)
  Interventions: Behavioral: Coping Together Booklets and Workbook; Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Coping Together Booklets and Workbook — Dyads in this group will complete Coping-Together, a 6-week, booklet-based, self-directed coping and self-management skills training intervention. This intervention addresses key psychosocial challenges by offering evidence-based practical skills to: (a) manage symptoms, (b) cope with anxiety, (c) collaborate with the health care team, (d) engage in shared decision-making, (e) communicate with partner and family, and/or (f) obtain the community resources needed. A relaxation CD is also included, in addition to a workbook that accompanies the Coping-Together booklet-based intervention. The workbook aims at helping dyads choose a booklet relevant to their cancer-related challenges faced, find coping skills that best meet these challenges, and make a plan to use one of the coping skills successfully.
Behavioral: Lay telephone coaching — Dyads will receive Coping-Together support via weekly telephone calls from a lay coach. Sessions will range between 10-15 minutes. The goal of coaching will be to provide information on how to use the workbook and booklets. Although no formal therapy will be provided, the coach will maintain a positive and encouraging attitude when interacting with participants regardless of their adherence to the intervention recommendations. The sessions will start with the coach setting a predetermined agenda based on the section of the workbook to review that week that week. Then, coaches will ask about the use of the booklets over the previous week, and ask participants about any required support or clarification in using the booklets. Sessions conclude with setting a goal related to the workbook, booklets and/or coping technique to focus on over the coming week.
  Arms: First stage: Minimally guided telephone support (lay coaching)
Behavioral: Motivational Interviewing — Six, 45-60 minute weekly telephone-based sessions with a trained Motivational Interviewing Specialist to progress toward goals. Here, dyads are given one-on-one guidance from a HCP Motivational Interviewing Specialist to practice the skills they need. Calls will focus on problem-solving principles and core components of self-management (70), including: (a) identifying dyads' concerns, (b) reviewing management efforts, (c) identifying goals, (d) identifying skills needed to achieve goals, and (e) addressing barriers to applying skills to current situations, including level of self-efficacy. At each meeting, progress, subsequent goals, and corresponding plans will be discussed.
  Arms: Second stage: High intensity Motivational Interviewing (MI)

SUMMARY:
High-quality cancer care in Canada relies on family caregivers. Since cancer treatment is provided more and more in outpatient clinics, family caregivers now provide most of the support and care patients need when they return home. The problem is that caregivers often do not feel they have the knowledge and skills to fulfill this role, especially as caregivers often confront tasks once performed by health care professionals. As a result, caregivers experience high levels of burden and need more help to handle the demands of their role. Programs that enhance caregivers' knowledge and prepare them for their role can have positive effects on their well-being. However, these programs are not available in routine cancer care. They just take too much time and personnel and are too expensive. This limited access to resources reduces caregivers' ability to cope and affects their quality of life. If the ultimate goal is to integrate these programs in cancer care, cost-effective service delivery models are needed. One approach that rises to this challenge and is effective is the self-directed format. A self-directed format requires less support from clinicians and is available to individuals when it is most convenient to them. The research team recently developed and evaluated the first self-directed coping skills training intervention for cancer caregivers called Coping-Together. Although self-directed interventions offer the scalability needed for public health interventions, up to 60% of caregivers do not improve after receiving this type of intervention. These caregivers require more support. This innovative trial design will help determine whether changing the type and level of support provided can increase the number of caregivers who improve after receiving Coping-Together. This type of innovative trial design is more and more popular, but has never been used to enhance the feasibility, acceptability, and efficacy of caregiver interventions.

DETAILED DESCRIPTION:
BACKGROUND: Despite improvements in detection and treatment, a cancer diagnosis is appraised as a negative event not only by the person diagnosed, but also by their family caregivers. Cancer is the second most common condition in Canada requiring assistance from caregivers, and caregivers are now taking on more than ever complex illness management roles traditionally performed by health care professionals (HCPs). This is in part attributed to the cost containment climate of the current health care system; there is an increased reliance on community-based care to manage the burden of cancer care on formal care settings. Caregivers' support reduces demands on the formal health care system and positively impacts on patients' adjustment. However, caregivers often take on their roles with little formal support. This results in high anxiety and low quality of life (QOL). In recognition of this, numerous interventions have been developed and found to be efficacious in reducing caregivers' anxiety and increasing their QOL. Unfortunately, these interventions are often time- and resource-intensive, making them too costly for integration in routine care. As more sustainable modes of intervention delivery are required, one format that holds promise is to use a self-directed format (i.e., low-intensity intervention). However, previous research by the team has shown that up to 60% of caregivers do not respond to these types of interventions alone and require additional support. An innovative trial design to developing time-varying, adaptive interventions to maximize clinical effectiveness is the Sequential multiple assignment randomized trials (SMARTs). However, despite increasing popularity, SMARTs remain relatively new to intervention researchers.

OBJECTIVES: The goal of this pilot SMART is to inform the planning of a subsequent larger SMART to evaluate an adaptive dyadic coping and self-management skill training intervention that follows a stepped-care model for caregivers of individuals with cancer. The primary objective of this pilot SMART is to examine the (a) feasibility of the trial procedures and of offering different levels and types of support alongside a self-directed coping and self-management skills training intervention and (b) acceptability of the combinations of the intervention according to patients and their caregivers. The secondary objective is to estimate the clinical significance of adapting the type and level of support provided on the primary and secondary outcomes.

METHODOLOGY: Study activities will be coordinated out of St Mary's Research Centre in Montreal. Weekly, at the McGill University Health Centre (MUHC), St. Mary's Hospital Center, and Ottawa Hospital, a research assistant (RA), along with the treating clinician, will screen new patient records and identify those who meet the medical inclusion criteria. At the time of their scheduled appointment, clinicians will introduce the study to eligible patients and obtain permission for a RA to approach them. The RA will then either complete the screening interview with patients and their caregivers on site, or follow up by telephone to complete the interview. Those eligible will be emailed the link to the consent form and baseline (T0) questionnaire. At BC Cancer Agency and Princess Margaret Cancer Care Centre, posters will be displayed and patients/caregivers will be informed of the study by the Patient and Family Counseling Services team and other health care team members. Patients will be invited to self-refer by calling the RA directly using the toll free number provided. Community-based recruitment will include advertising the study through social media. This strategy will be led by the Environics Research Group who recruited participants for a previous CIHR team grant.

Investigators aim to recruit 56 patients with a primary breast, prostate, or colorectal cancer diagnosis in the previous 6 months.

Inclusion criteria are:

* receiving/planning to receive treatment,
* having a caregiver willing to participate
* access to the internet,
* patient or caregiver screening positive for anxiety.

Patient-caregiver dyads returning their consent forms and baseline questionnaires (T0) will be randomized by the study coordinator to either: (a) Coping-Together - a 6-week self-directed, dyadic coping and self-management skills training intervention or (b) Coping-Together plus brief, weekly lay telephone coaching. At the end of 6 weeks, intervention response will be assessed by the RA (T1) based on the change in patients' and caregivers' anxiety (primary tailoring variable). Across both groups, non-responders will then be randomized a second time to either (a) continue with their first stage intervention or (b) begin telephone-based self-management counseling for another 6 weeks (either with a lay coach if self-directed for the first six weeks or with a health professional if coached for the first six weeks). Responders will continue with usual care. All participants will then complete their follow-up questionnaire (T2) to examine changes in anxiety and QOL (primary outcomes), depression, self-management skills, illness appraisal, and coping (secondary outcomes). Acceptability will also be assessed in this questionnaire and further explored during an exit interview with dyads. Feasibility measures will focus on the characteristics of the dyads reached, protocol fidelity, percent of missing data, and recruitment and retention rates.

SIGNIFICANCE: The ability of caregivers to maintain their QOL despite the stressors they face is undermined by limited access to the support needed. This study will develop and evaluate the first adaptive interventions for this population, and address a significant research gap by documenting its acceptability, feasibility, and clinical significance. Despite advocacy for caregiver support, no other Canadian study has examined how potentially cost-effective interventions can be combined to meet caregivers' needs. Collaboration with six cancer centers will accelerate the uptake of findings.

ELIGIBILITY:
Both patients with cancer and their caregivers will be recruited in this study as a dyad.

Inclusion Criteria:

* Stages I-III primary breast, prostate, or colorectal cancer diagnosis within the past 6 months
* receiving/planning to receive treatment (including surgery, radiotherapy, chemotherapy, and/or hormone therapy)
* nominates a caregiver (spouse, partner, or other family member) willing to participate
* patient and or caregiver with low-moderate anxiety at recruitment
* regular access to a computer with internet and e-mail capabilities,

Exclusion Criteria:

* caregiver receiving treatment for cancer
* patient or caregiver is hospitalized
* or has suicidal intent,
* or is receiving psychological treatment
* or has in the past 6 months participated in a coping or self-management program
* or has severe anxiety
* or has moderate-severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Consent and follow-up rates | From recruitment launch to completion of follow-up (9 months)
  Number of consenting dyads per week over the recruitment period, with report on refusal and drop-out rates and reasons.
Data completion rate | At T2: 13 weeks
  Investigators will report on rates of missing data from pilot baseline and follow-up questionnaires.
Fidelity of intervention delivery | At T2: 13 weeks
  Checklists will be used to assess if the interventions are delivered as per protocol
Adherence to intervention | At T2: 13 weeks
  Rate of tool use and participation in the support sessions.
Satisfaction with the intervention | At T2: 13 weeks
  Using a modified satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Hospital Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiesenfeld S, Lambert S, Laizner AM. A stepped-care approach to self-management: a qualitative study among individuals with cancer and their caregivers using the Coping-Together program. Support Care Cancer. 2025 Feb 10;33(3):170. doi: 10.1007/s00520-025-09175-5. PMID 39928172
- [Derived] Lambert S, Moodie EEM, McCusker J, Lokhorst M, Harris C, Langmuir T, Belzile E, Laizner AM, Brahim LO, Wasserman S, Chehayeb S, Vickers M, Duncan L, Esplen MJ, Maheu C, Howell D, de Raad M. Translating Evidence-Based Self-Management Interventions Using a Stepped-Care Approach for Patients With Cancer and Their Caregivers: A Pilot Sequential Multiple Assignment Randomized Trial Design. Psychooncology. 2025 Jan;34(1):e70043. doi: 10.1002/pon.70043. PMID 39763142